CLINICAL TRIAL: NCT05609747
Title: Effect of Non-Surgical Root Canal Treatment (NSRCT) on HbA1c and Inflammatory Markers in Healthy and Type 2 Diabetes Patients With Apical Periodontitis
Brief Title: Effect of NSRCT on HbA1c and Inflammatory Markers in Healthy and Type 2 Diabetes Patients With Apical Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Principal Investigator, Sanjay Tewari, HEAD OF THE DEPARTMENT, Postgraduate Institute of Dental Sciences Rohtak
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGIDS/BHRC/22/06/ NIKITA GARG
Record Dates: First submitted 2022-10-30; First posted 2022-11-08 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: PERIAPICAL LESIONS

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TYPE 2 DIABETIC PATIENTS (Experimental): NON SURGICAL ROOT CANAL TREATMENT
  Interventions: Procedure: Nonsurgical root canal therapy
- HEALTHY CONTROL GROUP PATIENTS (Experimental): NON SURGICAL ROOT CANAL TREATMENT
  Interventions: Procedure: Nonsurgical root canal therapy

INTERVENTIONS:
Procedure: Nonsurgical root canal therapy — After administration of LA and rubber dam isolation, acess cavity will be prepared using carbide burs in high speed hand piece with copious irrigation. Working length will be determined using root ZX apex locator and will be verified radiographically. Canal preparation will be done with protaper rotary instruments in which Sx to S2 will be used to shape the canals and F1 and F2 will be used to finish until the apex. 5ml of 5.25% NaOCl will be used as irrigant after each instrument. After instrumentation , the canals will be irrigated with 5.0 ml of 17% EDTA for 1minute followed by irrigation with 5.0 ml of 5.25% NaOCl. Canals will be dried with absorbent paper points, filled with calcium hydroxide paste and access cavity will be restored with IRM. Patients will be recalled after 1 week.At the next appointment, after paste removal, copious irrigation with 5.25% NaOCl will be done and canals will be dried with paper points. Canals will be obturated with Gutta-Percha and ZOE based sealer.
  Other Names: Root canal treatment

SUMMARY:
To the best of knowledge, only 2 prospective studies, and 1 cross-sectional study have been reported which have seen the periapical healing after non surgical endodontic treatment in diabetic patients and their effect on HbA1c.

Because of the inconsistencies in data available from the literature and considering the limitations of cross-sectional studies, further studies, especially using a prospective design, are required.

So, aim is to investigate the effects of non surgical endodontic treatment on healing and systemic inflammation in individuals with and without diabetes.

DETAILED DESCRIPTION:
Both the systematic review concluded that diabetics have significantly higher prevalence of RFT with RPL. An umbrella review concluded that DM is associated with the outcome of RCT and can be considered as a pre operative prognostic factor.

AP may contribute to low grade systemic inflammation associated with a generalized increase in systemic inflammatory mediators such as C-reactive protein (CRP), interleukin (IL)-1, IL-2, IL-6 and Immunoglobulin (IgA, IgG and IgM) levels .

It is already established that Diabetes mellitus (DM) and periodontitis are highly prevalent non-communicable diseases worldwide and yet they are closely inter-connected with common risk factors and plausibility of increased levels of systemic inflammation. It is evident that periodontitis significantly increases the risk of cardiovascular and renal complications in patients with type 2 diabetes mellitus (T2DM) . Higher serum high-sensitivity C-reactive protein (hsCRP) levels were reported in individuals with AP when compared to healthy controls . Also, there was a positive correlation of increased serum hsCRP levels with increasing severity of AP . A meta-analysis concluded that patients with AP had higher peripheral blood levels of CRP than controls and recommended the need for further studies to evaluate whether the treatment of AP can reduce serum CRP levels . Root canal treatment can reduce systemic inflammation and early endothelial dysfunction.

There is no published prospective interventional study evaluating the effect of root canal treatment on serum hsCRP levels in diabetic patients with AP.

Therefore, the aim of this study is to assess the impact of root canal treatment on HbA1c and serum hsCRP levels in diabetic adults with AP in comparison to healthy patients with AP.

ELIGIBILITY:
Inclusion Criteria:

* Known patient of type 2 diabetes mellitus with HbA1c ≥6.5 %. Age between 30 to 65 years. Mature permanent posterior tooth having apical periodontitis requiring primary root canal treatment.

No evidence of systemic diseases other than diabetes being a risk factor for apical periodontitis.

A radiographic evidence of periapical radiolucency (minimum size,≥2mm x2mm) and a diagnosis of pulpal necrosis, as confirmed by negative response to cold and electrical tests.

No antibiotic therapy within the preceding one month.

Exclusion Criteria:

* Teeth with procedural errors, cracks, fractured teeth. patients with previously endodontically treated teeth with periapical radiolucencies.

Teeth that were not suitable for rubber dam isolation. smokers, pregnant patients. Patients with moderate and severe periodontitis. Systemic diseases other than diabetes being a risk factor for apical periodontitis.

Immunocompromised patients.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2022-12-27 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Glycemic index (HbA1c) levels | Baseline to one year
  A hemoglobin A1C (HbA1C) test is a blood test that shows what your average blood sugar (glucose) level was over the past two to three months. A normal HbA1C level is below 5.7%, a level of 5.7% to 6.4% indicates prediabetes, and a level of 6.5% or more indicates diabetes
high sensitivity C- reactive protein- hsCRP. | Baseline to one year
  High-sensitivity C-reactive protein (hsCRP) (unit- mg/L)is a marker of inflammation that predicts incident myocardial infarction, stroke, peripheral arterial disease, and sudden cardiac death among healthy individuals with no history of cardiovascular disease, and recurrent events and death in patients with acute or stable coronary syndromes. hsCRP confers additional prognostic value at all levels of cholesterol, Framingham coronary risk score, severity of the metabolic syndrome, and blood pressure, and in those with and without subclinical atherosclerosis. hsCRP levels of less than 1, 1 to 3, and greater than 3 mg/L are associated with lower, moderate, and higher cardiovascular risks, respectively.

SECONDARY OUTCOMES:
Clinical and Radiographic success | Baseline to one year
  Absence of periapical alterations (radiolucency at furcal or periapical region) Scoring of each tooth will be done according to the following five point scale (PAI)
  Score Description
  1. Normal Periapical structure
  2. Small changes in bone structure
  3. Changes in bone structure with some mineral loss
  4. Periodontitis with well defined radiolucent area
  5. Severe periodontitis with exacerbating feature
  Lesions with a PAI score < 2 was considered as healed/healing.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - PGIDS, Rohtak, Haryana
  - Post Graduate Institute of Dental Science, Rohtak, Haryana

IPD SHARING:
Plan to Share IPD: No